CLINICAL TRIAL: NCT06861530
Title: A Swiss Prospective Multicenter Longitudinal Assessment of Hypothalamic-pituitary-adrenal Axis Suppression After Glucocorticoid Therapy for Leukemia and Lymphoblastic Lymphoma in Children: An Explorative Study
Brief Title: A Swiss Assessment of Hypothalamic-pituitary-adrenal Axis Suppression After Glucocorticoid Therapy for Leukemia and Lymphoblastic Lymphoma in Children
Acronym: LeukemiaCort
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00736
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Adrenal Insufficiency; Leukemia, Lymphoblastic, Acute, Pediatric; Lymphoma, Lymphoblastic
Keywords: Adrenal insufficiency; leukemia; leukaemia; childhood; pediatric; paediatric; glucocorticoid
MeSH Terms: conditions — Adrenal Insufficiency; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (Serum, EDTA)

GROUPS / COHORTS (1):
- Observed Cohort: Observed Cohort

SUMMARY:
Plain Language Summary:

Background Glucocorticoids are stress hormones produced by the human body to control inflammation and regulate the immune system. Cortisol is the most well-known example of a glucocorticoid. These stress hormones are essential for the bodys healthy functioning.

To treat certain types of cancer, such as leukemia (blood cancer) in children, glucocorticoids are administered as medications in large quantities. This helps rapidly reduce the number of cancer cells in the body but also leads to the suppression of the body's natural glucocorticoid production, causing a deficiency.

This deficiency can be particularly dangerous for children with leukemia, as their immune defenses are already weakened by chemotherapy, leading to an increased risk of infections. Moreover, the signs of glucocorticoid deficiency in children with leukemia are often indistinguishable from the side effects of chemotherapy, making the deficiency harder to detect.

Objectives The aim of the study is to understand how frequently and for how long the body's natural glucocorticoid production is impaired in children treated for lymphoblastic leukemia and lymphoblastic lymphoma. Additionally, the goal is to identify which children are at particularly high risk.

By gaining a better understanding, this study may help to improve the detection and treatment of glucocorticoid deficiency in children with blood cancer.

Methods Regular low-dose ACTH tests will be conducted to assess the bodys natural glucocorticoid production during and after treatment. To avoid placing additional burden on children who are already heavily affected by the disease, we will only perform these tests when there is already a venous access established and the children are in the hospital for treatment reasons.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ALL or LBL
* treated for at least 21 sequential days with glucocorticoids between the 01.07.2024 and the 30.06.2027 at the Childrens University Hospital of Basel or at the Childrens Hospital of Aarau
* lnformed consent can be obtained from the patient's legal representatives (and the patient if at least 14 years of age) within week 2 of treatment with glucocorticoids

Exclusion Criteria:

- Contraindication to the administration of intravenous synthetical ACTH (Synacthen®): extremely rare cases of known or suspected hypersensitivity to Synacthen®.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0-17 years who are:
  Diagnosed with ALL or LBL, and who are treated for at least 21 sequential days with glucocorticoids between the 01.07.2024 and the 30.06.2027 at the Childrens University Hospital of Basel or at the Childrens Hospital of Aarau
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurence of Adrenal Insufficiency | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  The primary outcome of this study is he measurement of the occurrence of HPA axis suppression. The outcome is binary (yes/no) and is considered yes, if a HPA axis suppression occurs at 1 test or more. HPA axis suppression is commonly defined as stimulated cortisol levels below 500nmol/l (below 18μg/dl) in the low-dose ACTH stimulation test, i.e. a measurement of cortisol 30 minutes and 60 minutes after the stimulation with 1 μg of synthetical ACTH (Synacthen®).
  For further analyses the following subgroups may be considered:
  - Morning cortisol according to current norm values from our laboratory: suppressed if below 66nmol/l (1-11 years) / below 100nmol/l (12-18 years)
  * Stimulated peak cortisol 300-500nmol/l = partially suppressed; below 300nmol/l = suppressed
  * Increment of cortisol after stimulation (basal to peak):
  below 100nmol/l = suppressed, 100-200nmol/l = partially suppressed, above 200nmol/l = normal

SECONDARY OUTCOMES:
Duration of Adrenal Insufficiency | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  The measurement of the duration of HPA axis suppression. The outcome is continuous (in weeks). lf there is no occurrence of HPA axis suppression (primary outcome, then this secondary outcome is 0 weeks.
  The cut-off values are specified under the primary outcome section.

OTHER OUTCOMES:
Number of infections | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  Number of infections: According to medical record. An infection is suspected at a temperature of at least 38.5°C (measured in hospital). This is a continuous outcome (in numbers).
Total days of hospitalization | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  Days of hospitalization: This is a continuous outcome (in numbers)
Total dose of glucocorticoid substitution | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  Total dose of glucocorticoid substitution: As decided by the treating physician. This is a continuous outcome (hydrocortisone in mg/m2/d)
Number of ICU admissions | Study enrollment until 3 months after the last dose of glucocorticoid treatment
  Number of ICU admissions. This is a continuous outcome (in numbers).

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - KSA, Aarau
  - UKBB, Basel

IPD SHARING:
Plan to Share IPD: No
not specified in approval by ethics comittee